CLINICAL TRIAL: NCT00481624
Title: A Phase II Trial Using Intravenous Iron in Advanced Lung Cancer Patients With Chemotherapy-Induced Anemia Treated With 120,000 Units Epoetin Alfa Every Three Weeks
Brief Title: Using Iron With Procrit in Advanced Lung Cancer Patients With Chemotherapy-Induced Anemia
Acronym: Procrit
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped because of lack of funding.
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Goetz Kloecker, Associate Professor, University of Louisville
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07.0210
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Anemia
Keywords: advanced lung cancer; Procrit; Epoetin Alfa; Ferric Gluconate; iron supplementation
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa; Iron; ferric gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epoetin Alfa plus Iron (Experimental)
  Interventions: Drug: Epoetin Alfa plus Iron

INTERVENTIONS:
Drug: Epoetin Alfa plus Iron — 1. One (1) injection of Procrit®, by needle, inserted just under the skin;
  2. 125 mg of ferric gluconate (an iron injection product), through an IV injection into a vein.
  These injections will take approximately 10-15 minutes to complete. Both will be administered every 3 weeks for a total of 4 cycles, unless the study doctor decides that a change in the amount of Procrit® and iron is necessary once the hemoglobin level rises or is above a certain amount.
  In addition to Procrit® and the intravenous iron, the subject will also receive platinum-containing chemotherapy every 3 weeks for 4 cycles as per standard of care for their lung cancer treatment. Radiation therapy will be allowed during this regimen if it is part of the subject's treatment plan.
  Other Names: Procrit®; Ferrlecit®

SUMMARY:
The purpose of this study is to find a better, more convenient way to improve anemia results by increasing the amount of medication given at 3 week intervals. Researchers want to know if giving a higher dose of Procrit® and intravenous (IV) iron once every 3 weeks would give better results in treating anemia without the need for more office visits.

DETAILED DESCRIPTION:
There are more than 170,000 patients diagnosed with lung cancer in the United States each year and many will develop anemia (iron deficiency) during the course of treatment. Anemia is associated with poor quality of life and treatment delays for advanced lung cancer. The treatment of iron deficiency anemia is with iron. Iron is an essential mineral used in red blood cells to carry oxygen throughout the body. Iron is necessary to make hemoglobin, a key element in red blood cells.

The FDA has approved Procrit® (epoetin alfa) to treat anemia in people with non-myeloid (bone marrow) malignancies. Procrit® is a man-made, injectable drug for treating anemia and it encourages red cell production. While the administration of intravenous iron therapy, injected into veins through an IV, did increase the response rate of Procrit® in a previous study, researchers want to find out the best amount of drug to use and the best time to administer Procrit®, along with ferric gluconate, (Ferrlecit®), added for lack of iron.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed small cell or non small cell lung cancer
* Stage III or Stage IV lung cancer
* Platinum containing chemotherapy induced anemia (< 10 g/dl Hb)
* Cancer related anemia (<10 g/dl Hb) at time of initiation of chemotherapy
* ECOG performance status of 0,1, or 2
* Informed consent
* Age>18
* Expected to receive platinum based outpatient chemotherapy for at least nine weeks

Exclusion Criteria:

* Pregnant women
* Intolerance to epoetin alfa or parenteral iron
* More than 2 cycles of the planned platinum chemotherapy at time of enrollment
* Chronic GI bleed (> than 4 weeks positive hemoccult or gastroccult)
* Ferritin > 500 mg/dl
* Anemia due to other causes than cancer or chemotherapy
* Previous parenteral iron therapy
* Uncontrolled hypertension (systolic BP > 160, diastolic > 100 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Achieve hemoglobin responses > 2g/dl in at least 70% of patients | Nine weeks, after at least two doses of 120,000 units epoetin alfa

SECONDARY OUTCOMES:
Descriptive evaluation of adverse effects of parenteral iron and epoetin alfa 120,000 units given every three weeks | Patient follow up until week 12

CONTACTS AND LOCATIONS:
Overall Officials: Goetz H Kloecker, MD, Principal Investigator — James Graham Brown Cancer Center, Univeristy of Louisville
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

REFERENCES:
- See also: James Graham Brown Cancer Center, Louisville, KY — http://www.browncancercenter.org